CLINICAL TRIAL: NCT07151976
Title: Pathologic Features of Aspirated Athero-Thrombotic Material From OCT-Verified Culprit Lesion in Acute Coronary Syndrome (TAPOS)
Brief Title: Thrombus Aspiration and Pathology and OCT Study
Acronym: TAPOS
Status: Recruiting | Type: Observational
Sponsor: Fujita Health University (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Yukio Ozaki, Clinical Professor, Fujita Health University
Other Study IDs: HM22-157
Record Dates: First submitted 2022-02-10; First posted 2025-09-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Human atherosclerotic material
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PCI — PCI with athero-thrombotic aspiration and subsequent pathological analysis: Pathologic Characteristics of Athero-Thrombotic AsPirated Material of OCT-Verified Culprit Lesion in Acute Coronary Syndrome

SUMMARY:
Most acute coronary syndromes (ACS) are caused by plaque complications triggering thrombotic events in the culprit plaques. Plaque complications include plaque rupture (Ruptured Fibrous Cap-RFC) with exposure of highly thrombogenic substrate to the flow and plaque erosion (Intact Fibrous Cap-IFC) a condition characterized by endothelial/intimal damage occurring over non-ruptured plaques. Far less commonly (<5%), calcified nodules (CN) may trigger acute coronary thrombosis. Plaque rupture accounts for 75% of fatal AMI in autopsy series, while erosion is found in about 25% of cases. These proportions have been supported by in vivo invasive studies (OCT) and OCT-pathology correlation studies. However, it remains unclear whether OCT findings consistently align with in vivo pathology-based evidence of RFC in ACS. Guidelines addressing treatments of ACS unanimously indicate percutaneous coronary intervention (PCI) to restore the coronary flow. Pre-PCI thrombus aspiration is not currently indicated by most guidelines, with the exception of cases with very high thrombus burden. The samples retrieved from thrombus aspiration can be suitable for pathology investigation and aim to evaluate the presence of plaque components in the context of the thrombotic material, a finding that demonstrates plaque rupture as the substrate for the acute coronary event. These studies are uniquely qualified to provide information on the correct OCT-based interpretation of plaque complications in ACS and require OCT imaging quality suitable to classify RFC, IFC, and CN.

Therefore, a prospective OCT-pathology study was designed using the pre-PCI aspirated material from patients with high thrombus burden, to explore the contribution of pathology study in OCT-based classification of plaque complications.

DETAILED DESCRIPTION:
AIM Primary aim The present study aims to assess whether the composition of thrombus-aspirated material differs in samples retrieved from patients with OCT-described plaque rupture, erosion, or calcified nodules. In particular, the specific aim is to assess the presence of plaque components (atheromatous material, consisting of cholesterol clefts, foam cells, iron-loaded macrophages, cap fragments, and calcifications) in plaques described at OCT as RFC, IFC, and CN. The working hypothesis is that the pre-PCI aspirated material from plaque rupture should contain plaque components, while aspirated material from plaque erosion, should only contain thrombotic material. The pathology study was planned to be performed blindly to imaging data, and report independent descriptors of the pathology features.

Secondary aims

1. A secondary aim addresses pathophysiology mechanisms, potentially related to features promoting plaque rupture. Given the proposed major role of macrophages in the context of plaque inflammation commonly observed in vulnerable plaque prone to rupture, we aimed to investigate the presence of M1 (pro-inflammatory, pro-rupture effect) and M2 (anti-inflammatory, anti-rupture effect) macrophages in samples containing plaque material.
2. A further secondary aim is the assessment of short- and long-term outcomes in patients with OCT-diagnosed plaque complications, as identified by imaging and confirmed by pathology.

SAMPLE SIZE Due to the unprecedented similar in vivo studies and the non-routine possibility of performing pre-PCI thrombus aspiration according to guidelines, it was not possible to precisely calculate the sample size.

Based on the probability of plaque rupture in ACS (75% in consecutive ACS) and erosion (25% in consecutive series), a minimum number of 100 cases was considered necessary for the study scope.

PATIENT RECRUITMENT The study is conducted at the Fujita Health University Hospital, Okazaki Medical Center, and Nagoya First Red Cross Hospital. The study was approved by local ethics committees (HM 16019) and was carried out according to the guidelines of the Declaration of Helsinki. Written informed consent was obtained from all patients before index PCI.

PATHOLOGICAL ANALYSIS The pathologic study was planned to be performed at the IRCCS, Policlinico San Matteo, Pavia, Italy, where samples had to be blindly analyzed after routinely processing for histopathology.

Pathological plaque rupture (PATHO-PR) was defined as the presence within the retrieved samples of atheromatous material, consisting of cholesterol clefts, foam cells, iron-loaded macrophages, cap fragments/fibrous tissue, and calcifications.

Serial sections for each case were stained (H&E, MOVAT, Perls', Von Kossa). The immuno-characterization of the macrophage populations was performed by immunostaining sample sections with antibodies to the pan-macrophage CD68, and M1 (CD80, CD86, IL-6) and M2 (CD163, CD206, TGF-β) polarized macrophage.

Samples with plaque material were classified as RFC-derived, while thrombus-only samples were unsuitable for plaque analysis.

CLINICAL EVALUATION Clinical outcomes were planned at 100 days and 5 years. Major adverse cardiac events (MACE) included cardiac death, non-fatal ACS, ischemia-driven revascularization, cardiogenic shock, and heart failure requiring hospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ACS showing ST-segment elevation myocardial infarction (STEMI) or non-ST-segment elevation myocardial infarction (NSTEMI) are studied.
2. Only native coronary artery lesions are included in the study.
3. Optical coherence tomography (OCT) was performed prospectively to compare OCT culprit lesions characteristics with histological analysis of athero-thrombotic aspirated material of the culprit lesion. For this purpose, only lesions with both athero-thrombotic aspirated material and OCT observations are included in the study.
4. All patients provided written informed consent for the index procedure, follow-up, and anonymous data management.

Exclusion Criteria:

1. Patients are excluded from the study when they had cardiogenic shock and contraindications to anticoagulation and anti-platelet therapy.
2. Lesions located in tortuous vessels, in ostial segment and in the left main stem are excluded from the study due to the difficulty in performing high-quality intracoronary imaging.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between July 2016 and December 2024, 200 consecutive patients with ACS having large angiographic thrombus burden who assumed to have a merit of thrombotic aspiration and who consented to OCT guided PCI procedures with athero-thrombotic aspiration were enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Concordance between pathology based and optical coherence tomography (OCT) verified diagnosis of plaque rupture | From 2016 to 2027
  TAPOS is an observational prospective study that aims to investigate the concordance between pathology versus OCT-verified features of plaque rupture in patients with STEMI and NSTEMI undergoing PCI and athero-thombus aspiration from the culprit coronary plaque. Pathology measured features are assessed in the aspirated material retrieved from the target coronary plaque and include the presence of foam or iron-loaded macrophages, cholesterol clefts, fragments of fibrous tissue, and calcifications assessed as single or combined features. OCT-based features of plaque include coronary thrombi, fibrous cap discontinuity or plaque ulceration (contraposed to non-ruptured, continuous fibrous cap with over-imposed thrombus).

SECONDARY OUTCOMES:
Concordance between pathology-based and optical coherence tomography (OCT) verified detection of macrophages | From 2016 to 2027
  TAPOS is an observational prospective study that investigates the concordance between pathology vs. OCT-verified features of plaque rupture in patients with STEMI and NSTEMI undergoing PCI and thrombus aspiration from the culprit coronary plaque. Pathology measured features assessed in the aspirated material retrieved from the target coronary plaque include the presence of foam- or iron-loaded macrophages, cholesterol clefts, fragments of fibrous tissue, and calcifications, as single or combined feature/s. OCT-based features of plaque rupture include fibrous cap discontinuity, plaque ulceration (contraposed to non-ruptured, continuous fibrous cap with over-imposed thrombus).
  In addition, TAPOS investigates the correlation between the OCT-based detection of macrophages (signal-rich, distinct, or confluent punctate regions that exceed the intensity of background speckle noise) and the pathology observation of macrophages in the thrombus-aspirated material retrieved from each lesion.
The incidence rate of major adverse cardiac events (MACE) | From 2016 to 2027
  Major adverse cardiac and cerebral events (MACE): the composite of cardiac death, non-fetal MI, and unstable angina requiring PCI or CABG
The incidence rate of major adverse cardiac and cerebrovascular events (MACCE) | From 2016 to 2027
  Major adverse cardiac and cerebral events (MACCE): the composite of cardiac death, non-fetal MI, and unstable angina requiring PCI or CABG, and stroke
The incidence rate of major adverse cardiac and fatal events | From 2016 to 2027
  Major adverse cardiac and cerebral events: the composite of all-cause death, non-fetal MI, and unstable angina requiring PCI or CABG
The incidence rate of major cardiac, cerebrovascular, and fatal events | From 2016 to 2027
  Major adverse cardiac and cerebral events: the composite of all-cause death, non-fetal MI, and unstable angina requiring PCI or CABG, and stroke

CONTACTS AND LOCATIONS:
Overall Officials: YUKIO OZAKI, MD, PhD, Principal Investigator — Fujita Health University, Aichi, Japan; Eloisa Arbustini, MD, Study Chair — IRCCS Foundation Policlinico San Matteo, Pavia, Italy
Locations (1):
- Fujita Health University, Toyoake, Aichi-ken, Japan